CLINICAL TRIAL: NCT07373886
Title: Suprapubic Transverse Incision With Rectus Release for Upper Peritoneal Access): A Novel Dual-Plane Technique for Abdominal Wall Incision in Complex Gynecological Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdalla Mousa, Lecturer of Obstetrics and Gynecology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MS-599-2025
Record Dates: First submitted 2026-01-21; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Post-Op Complication
MeSH Terms: conditions — Postoperative Complications | interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STIRRUP (Suprapubic Transverse Incision with Rectus Release for Upper Peritoneal access) technique (Experimental): Skin incision: A low curvilinear transverse incision will be made 2-3 cm above the pubic symphysis, corresponding to the Pfannenstiel site.
  Subcutaneous dissection: The subcutaneous tissue will be elevated between Scarpa's fascia and the anterior rectus sheath for approximately 10-12 cm cephalad.
  Anterior rectus sheath incision: A transverse incision will be made in the anterior rectus sheath approximately 10-12 cm above the pubis, parallel to the skin incision. The linea alba will not be divided, thereby preserving midline fascial integrity.
  Rectus muscle separation: Beneath the fascial window, the rectus muscles will be separated bluntly at the midline, as in the Pfannenstiel approach, to expose the posterior sheath and peritoneum. No transection of muscle fibers will be performed.
  Peritoneal entry: The peritoneum will be opened sharply under direct vision.
  Interventions: Procedure: STIRRUP (Suprapubic Transverse Incision with Rectus Release for Upper Peritoneal access) technique

INTERVENTIONS:
Procedure: STIRRUP (Suprapubic Transverse Incision with Rectus Release for Upper Peritoneal access) technique — Skin incision: A low curvilinear transverse incision will be made 2-3 cm above the pubic symphysis, corresponding to the Pfannenstiel site.
  Subcutaneous dissection: The subcutaneous tissue will be elevated between Scarpa's fascia and the anterior rectus sheath for approximately 10-12 cm cephalad.
  Anterior rectus sheath incision: A transverse incision will be made in the anterior rectus sheath approximately 10-12 cm above the pubis, parallel to the skin incision. The linea alba will not be divided, thereby preserving midline fascial integrity.
  Rectus muscle separation: Beneath the fascial window, the rectus muscles will be separated bluntly at the midline, as in the Pfannenstiel approach, to expose the posterior sheath and peritoneum. No transection of muscle fibers will be performed.
  Peritoneal entry: The peritoneum will be opened sharply under direct vision.

SUMMARY:
This study aims to evaluate the clinical effectiveness, anatomical benefits, and postoperative outcomes of the STIRRUP incision (Suprapubic Transverse Incision with Rectus Release for Upper Peritoneal Access) by comparing outcomes with historically established benchmarks and published data from traditional abdominal wall incisions used in complex gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-65 years
2. Indication for open gynecologic surgery for benign or borderline pelvic or abdominopelvic masses
3. Body Mass Index (BMI) ≥ 18 kg/m²
4. Willing and able to provide informed consent and attend follow-up
5. Mass size between 15-30 cm, which is considered optimal for the STIRRUP (Suprapubic Transverse Incision with Rectus Release for Upper Peritoneal access) technique due to the balance between exposure and minimal morbidity

Exclusion Criteria:

1. Malignant tumors requiring upper abdominal visceral resection (liver, spleen, diaphragm)
2. Emergency surgery
3. Previous complex abdominal wall reconstruction with mesh
4. Contraindication to general anesthesia
5. Masses extending to the xiphisternum or measuring >30 cm
6. Cases requiring supracolic omentectomy
7. Planned lymphadenectomy (especially if comprehensive para-aortic lymph node dissection is required )
8. Supramesocolic tumor extension or malignant ovarian tumors requiring hepatic resections, splenectomy, and diaphragmatic resection
9. Severe comorbidities precluding elective surgery
10. Pregnancy
11. Previous extensive upper abdominal surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative seroma formation | within the postoperative or follow-up period (6 months)
  clinically detectable subcutaneous fluid collection at the incision site, confirmed clinically and/or by ultrasound when indicated.